CLINICAL TRIAL: NCT04719000
Title: PErsonalized Addition of Recombinant LH in Suboptimal Responders >35 Years Old (POSEIDON Group 2): A Randomized Controlled Trial
Brief Title: PErsonalized Addition of Recombinant LH in Ovarian Stimulation
Acronym: PEARL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Santiago Dexeus Font (Other)
Collaborators: Merck, S.L., Spain (Industry)
Responsible Party: Sponsor
Organization: Fundacion Dexeus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FSD-RHLH-2019-08
Record Dates: First submitted 2021-01-14; First posted 2021-01-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rhFSH+rhLH (Experimental): Ovarian Stimulation with rhFSH+rhLH
  Interventions: Drug: rhFSH+rhLH
- rhFSH (Active Comparator): Ovarian Stimulation with rhFSH
  Interventions: Drug: rhFSH

INTERVENTIONS:
Drug: rhFSH+rhLH — 300 IU of rhFSH and 150 IU of rhLH (Pergoveris®) GnRH antagonist: cetrorelix 0.25 mg (Cetrotide® - Merck) GnRH antagonist: cetrorelix 0.25 mg (Cetrotide® - Merck) Recombinant human chorionic gonadotropin (rhCG) 6500 IU (Ovitrelle® - Merck) micronized progesterone 90 mg (Crinone 8% ® - Merck)
  Arms: rhFSH+rhLH
Drug: rhFSH — 300 IU rhFSH (Gonal-F®- Merck) GnRH antagonist: cetrorelix 0.25 mg (Cetrotide® - Merck) GnRH antagonist: cetrorelix 0.25 mg (Cetrotide® - Merck) rhCG 6500 IU (Ovitrelle® - Merck) micronized progesterone 90 mg (Crinone 8% ® - Merck)
  Arms: rhFSH

SUMMARY:
Different ovarian stimulation regimens have shown to modify late follicular phase hormonal profiles. Besides, recent studies confirm that progesterone levels and their variation in the last day of oocyte maturation are affected by the dose of gonadotropins administered and by other factors. Progesterone elevation in late follicular phase of in vitro fertilization/intracytoplasmatic sperm injection (IVF/ICSI) cycles under ovarian stimulation compromises implantation rates due to a negative effect on the endometrium. However, there is still conflict in the literature questioning whether progesterone levels alone on the triggering day is a sufficient indicator as progesterone does not give the full picture of the ovarian functions, number of follicles as well as estrogen production that facilitate endometrial growth, thus some studies suggest that especially in aged and poor responders Progesterone/Estrogen (P4/E2) ratio has a better reflection (Progesterone (ng/mL) ×1,000/estradiol(pg/mL)) on the ovarian function.

The scope of the current pilot study is to compare serum progesterone levels as well as P4/E2 ratio on the day of ovulation triggering of women belonging to POSEIDON category group 2 who undergo a new ovarian stimulation with a dose of rhFSH 300 IU or 300 IU rhFSH plus 150 IU recombinant human luteinizing hormone (rhLH) in a gonadotropin-releasing hormone (GnRH) antagonist protocol.

DETAILED DESCRIPTION:
The main objective of assisted reproductive technology is to achieve a healthy child. Many aspects play a role in order to reach this outcome, including female age, the number of oocytes retrieved after ovarian stimulation, and endometrial receptivity. It has been clearly demonstrated that the number of oocytes obtained after ovarian stimulation for IVF/ICSI is a surrogate marker for the success rates following treatment. In general, a high number of oocytes retrieved is translated into a high number of embryos and eventually a high cumulative pregnancy rate (after the transfer of fresh and frozen-thawed embryos). However, although a higher number of oocytes and embryos may ensure an increase in the cumulative pregnancy rate, excessive ovarian response has been postulated to have a detrimental effect on the pregnancy rates following fresh embryo transfer given that raised serum estradiol and progesterone levels associated with a very excessive response may negatively affect embryo implantation.

In assisted reproductive technology (ART) cycles under the GnRH analog regimens, elevated progesterone serum levels at the late follicular phase, in good ovarian reserve women, is thought to be related to multiple follicular development and increased ovarian steroidogenic activity. However, for these patients elevated progesterone was shown to negatively affect the endometrium preparation and thereby implantation rate. Furthermore, in this group of women elevated progesterone is advocated to have no negative effect on the oocyte or embryo quality.

Importantly, more pronounced effect on unbalanced steroidogenesis has been correlated with age and ovarian reserve. For this patient population, serum progesterone/estradiol (P/E2) ratio on the day of human chorionic gonadotropin (hCG) administration was suggested as a more reliable marker predictor to cycle success than solely progesterone rise.

Based on the above-mentioned reports it is relatively clear that the aim of ovarian stimulation should be to result in high oocyte yield and educate endocrine milieu in order to maximize cumulative live birth rates. Nevertheless, despite this goal, a substantial proportion of patients do not manage to reach an optimal oocyte yield, resulting in lower pregnancy rates. These hypo-responders are associated with low follicles growth and reduced estrogen production leading to longer stimulations, and/or greater cumulative FSH doses.

Although, it is widely accepted that poor ovarian responders have significantly low live birth rates as compared with all other groups, an intermediate group of women with a "suboptimal ovarian response", has been recently proposed as a distinct group with significantly worse prognosis from women with normal response. In the same line, the POSEIDON group (Patient-Oriented Strategies Encompassing IndividualizeD Oocyte Number) has recently proposed a new stratification for patients with a reduced ovarian reserve or unexpected inappropriate ovarian response to ovarian stimulation, taken into account quantitative and qualitative parameters such as: i. Age and the expected aneuploidy rate; ii. Ovarian biomarkers (mainly antral follicle count (AFC) and anti-Müllerian hormone (AMH)), and iii. Ovarian response to a previous stimulation cycle.

One of the most interesting group of patients fulfilling the POSEIDON criteria is undeniably, POSEIDON GROUP 2: Women ≥35 years with adequate ovarian reserve parameters (AFC≥5; AMH≥1.2 ng/ml) and with unexpected poor or suboptimal ovarian response:

* Subgroup 2a: <4 oocytes after standard ovarian stimulation.
* Subgroup 2b: 4-9 oocytes after standard ovarian stimulation.

Patients belonging to the POSEIDON group 2 are women with an objectively good ovarian reserve who do not manage to respond as expected following ovarian stimulation. Consequently, taking into account that these patients are women who do not respond in accordance to their ovarian reserve following ovarian stimulation, identifying the optimal treatment protocol for these women remains of paramount importance, namely these patients show slow response to FSH stimulation in terms of estradiol levels and follicle growth, require longer stimulations, and/or greater cumulative FSH doses despite their correct ovarian parameters.

In this regard, different gonadotropins used for ovarian stimulation have shown to affect differently late follicular phase hormonal levels. In fact, although the role of LH in the follicular phase of ovarian stimulation is still a matter of debate, it seems that IVF/ICSI cycles under LH activity reach lower progesterone levels on the day of ovulation triggering. However, no study has evaluated late follicular phase progesterone levels in Poseidon 2 group patients receiving recombinant FSH (rhFSH) versus rhFSH and rhLH for ovarian stimulation.

Taking into account the above-mentioned evidence, the investigators set out to perform a pilot study in women with suboptimal response (fulfilling Poseidon 2 criteria), in order to examine whether the addition of rhLH to rhFSH significantly changes late follicular phase progesterone levels as compared to rhFSH alone.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to sign the Patient Consent Form and adhere to study visitation schedule.
* ≥ 35 years ≤40 years old.
* AFC ≥5 and or AMH ≥1.2 ng/mL.
* <4 or 4-9 oocytes retrieved in a previous IVF/ICSI cycle with a starting dose of ≤225 IU with any gonadotropin under a GnRH antagonist protocol.
* Up to 3 previous ovarian stimulation cycles with a starting dose of ≤225 IU in which dose adjustments during stimulation did not exceed 300 IU.
* Ovarian stimulation for IVF/ICSI

Exclusion Criteria:

* Poor ovarian responders according to the Bologna criteria.
* Polycystic ovary syndrome (PCOS) patients according to the Rotterdam criteria.
* AFC>20.
* Age >40 or <35 years old.
* Women with >10 oocytes retrieved in a previous IVF/ICSI cycle with 150-225 IU starting dose.
* Women who required dose adjustments during stimulation >300 IU with any gonadotropin in their previous cycle
* Uterine abnormalities.
* Recent history of any current untreated endocrine abnormality.
* Unilateral or bilateral hydrosalpinx (visible on ultrasound scan (USS), unless clipped).
* Contraindications for the use of medicine used for ovarian stimulation (gonadotropins, GnRH antagonist, progesterone vaginal gel)
* Recent history of severe disease requiring regular treatment (Clinically significant concurrent medical condition that could compromise subject safety or interfered with the trial assessment and patients with any contraindication to pregnancy).
* Preimplantation Genetic Testing for Aneuploidies (PGT-a).
* Testicular Sperm Aspiration or Testicular Sperm Extraction (TESA or TESE)

Ages: 35 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-02-04 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Serum progesterone levels on the day of ovulation triggering. | 5 -20 days from initiation of ovarian stimulation
  The outcome will be evaluated on the day of ovulation triggering
P/E2 ratio | 5 -20 days from initiation of ovarian stimulation
  Progesterone / estradiol ratio

SECONDARY OUTCOMES:
Progesterone Profile | days 1, 6, 8, 10 and the day of ovulation triggering
Estradiol Profile | days 1, 6, 8, 10 and the day of ovulation triggering
FSH Profile | days 1, 6, 8, 10 and the day of ovulation triggering
Testosterone Profile | days 1, 6, 8, 10 and the day of ovulation triggering
LH Profile | days 1, 6, 8, 10 and the day of ovulation triggering
P/E2 ratio Profile | days 1, 6, 8, 10 and the day of ovulation triggering
Values of Progesterone-to-follicle Index (PFI) | on the day of ovulation triggering.
Oocytes retrieved | 7 -20 days from initiation of ovarian stimulation
Metaphase II (MII) oocytes retrieved | 7 -20 days from initiation of ovarian stimulation
Follicle to Oocyte Indexs (FOI) | 7 -20 days from initiation of ovarian stimulation
  ratio between the total number of oocytes collected at the end of ovarian stimulation and the number of antral follicles available at the start of stimulation
Follicular Output Rates (FORT) | Day 1 at the start of stimulation
  ratio of the number of preovulatory follicles and the number of antral follicles available at the start of stimulation
Percentage of patients with optimal number of oocytes retrieved (≥10 oocytes). | 7 -20 days from initiation of ovarian stimulation
Percentage (%) of top-quality embryos | Until 5, 6 or 7 days after insemination
Blastocyst formation rates (%). | Until 5, 6 or 7 days after insemination
Clinical pregnancy | at 6-7 weeks of gestation
  defined as the presence of intrauterine gestational sac with an embryonic pole demonstrating cardiac activity
Ongoing pregnancy | at 8-9 weeks of gestation
  defined as the presence of intrauterine gestational sac with an embryonic pole demonstrating cardiac activity
Biochemical pregnancy | 2 weeks after embryo transfer
  defined as positive pregnancy test

OTHER OUTCOMES:
Ovarian hyperstimulation syndrome (OHSS) (percent). | Until 15 days after the end of ovarian stimulation
  Number of subjects with OHSS during the ovarian stimulation period and their severity
Miscarriages | before completion of 12 weeks of gestation
  any spontaneous abortion that occurred after confirmation of clinical pregnancy
Cycle cancelation | Until 15 days after the beginning of ovarian stimulation
  when no follicle has adequate maturation or the follicle is lost due to spontaneous LH surge
Incidence of adverse events and serious adverse events | Until 15 days after the end of ovarian stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos P Polyzos, MD PhD, Study Chair — Hospital Universitari Dexeus
Locations (1):
- Hospital Universitario Quiron Dexeus, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Esteves SC, Khastgir G, Shah J, Murdia K, Gupta SM, Rao DG, Dash S, Ingale K, Patil M, Moideen K, Thakor P, Dewda P. Association Between Progesterone Elevation on the Day of Human Chronic Gonadotropin Trigger and Pregnancy Outcomes After Fresh Embryo Transfer in In Vitro Fertilization/Intracytoplasmic Sperm Injection Cycles. Front Endocrinol (Lausanne). 2018 Apr 26;9:201. doi: 10.3389/fendo.2018.00201. eCollection 2018. PMID 29755412
- [Background] Fatemi HM, Van Vaerenbergh I. Significance of premature progesterone rise in IVF. Curr Opin Obstet Gynecol. 2015 Jun;27(3):242-8. doi: 10.1097/GCO.0000000000000172. PMID 25811257
- [Background] Huang Y, Wang EY, Du QY, Xiong YJ, Guo XY, Yu YP, Sun YP. Progesterone elevation on the day of human chorionic gonadotropin administration adversely affects the outcome of IVF with transferred embryos at different developmental stages. Reprod Biol Endocrinol. 2015 Aug 4;13:82. doi: 10.1186/s12958-015-0075-3. PMID 26238449
- [Background] Joo BS, Park SH, An BM, Kim KS, Moon SE, Moon HS. Serum estradiol levels during controlled ovarian hyperstimulation influence the pregnancy outcome of in vitro fertilization in a concentration-dependent manner. Fertil Steril. 2010 Feb;93(2):442-6. doi: 10.1016/j.fertnstert.2009.02.066. Epub 2009 Apr 25. PMID 19394001
- [Background] Lawrenz B, Fatemi HM. Effect of progesterone elevation in follicular phase of IVF-cycles on the endometrial receptivity. Reprod Biomed Online. 2017 Apr;34(4):422-428. doi: 10.1016/j.rbmo.2017.01.011. Epub 2017 Jan 24. PMID 28162937
- [Background] Mitwally MF, Bhakoo HS, Crickard K, Sullivan MW, Batt RE, Yeh J. Estradiol production during controlled ovarian hyperstimulation correlates with treatment outcome in women undergoing in vitro fertilization-embryo transfer. Fertil Steril. 2006 Sep;86(3):588-96. doi: 10.1016/j.fertnstert.2006.02.086. Epub 2006 Jun 30. PMID 16814289
- [Background] Valbuena D, Martin J, de Pablo JL, Remohi J, Pellicer A, Simon C. Increasing levels of estradiol are deleterious to embryonic implantation because they directly affect the embryo. Fertil Steril. 2001 Nov;76(5):962-8. doi: 10.1016/s0015-0282(01)02018-0. PMID 11704118
- [Background] Racca A, De Munck N, Santos-Ribeiro S, Drakopoulos P, Errazuriz J, Galvao A, Popovic-Todorovic B, Mackens S, De Vos M, Verheyen G, Tournaye H, Blockeel C. Do we need to measure progesterone in oocyte donation cycles? A retrospective analysis evaluating cumulative live birth rates and embryo quality. Hum Reprod. 2020 Jan 1;35(1):167-174. doi: 10.1093/humrep/dez238. PMID 31953546
- [Background] Younis JS. The role of progesterone/estradiol ratio in exploring the mechanism of late follicular progesterone elevation in low ovarian reserve women. Med Hypotheses. 2019 Apr;125:126-128. doi: 10.1016/j.mehy.2019.02.047. Epub 2019 Feb 28. PMID 30902140
- [Background] Lin YJ, Lan KC, Huang FJ, Lin PY, Chiang HJ, Kung FT. Reproducibility and clinical significance of pre-ovulatory serum progesterone level and progesterone/estradiol ratio on the day of human chorionic gonadotropin administration in infertile women undergoing repeated in vitro fertilization cycles. Reprod Biol Endocrinol. 2015 May 13;13:41. doi: 10.1186/s12958-015-0037-9. PMID 25967104
- [Background] Grynberg M, Labrosse J. Understanding Follicular Output Rate (FORT) and its Implications for POSEIDON Criteria. Front Endocrinol (Lausanne). 2019 Apr 16;10:246. doi: 10.3389/fendo.2019.00246. eCollection 2019. PMID 31040828
- [Background] Polyzos NP, Nwoye M, Corona R, Blockeel C, Stoop D, Haentjens P, Camus M, Tournaye H. Live birth rates in Bologna poor responders treated with ovarian stimulation for IVF/ICSI. Reprod Biomed Online. 2014 Apr;28(4):469-74. doi: 10.1016/j.rbmo.2013.11.010. Epub 2013 Dec 4. PMID 24581984
- [Background] Polyzos NP, Sunkara SK. Sub-optimal responders following controlled ovarian stimulation: an overlooked group? Hum Reprod. 2015 Sep;30(9):2005-8. doi: 10.1093/humrep/dev149. Epub 2015 Jul 21. PMID 26202582
- [Background] Sunkara SK, Rittenberg V, Raine-Fenning N, Bhattacharya S, Zamora J, Coomarasamy A. Association between the number of eggs and live birth in IVF treatment: an analysis of 400 135 treatment cycles. Hum Reprod. 2011 Jul;26(7):1768-74. doi: 10.1093/humrep/der106. Epub 2011 May 10. PMID 21558332
- [Background] Poseidon Group (Patient-Oriented Strategies Encompassing IndividualizeD Oocyte Number); Alviggi C, Andersen CY, Buehler K, Conforti A, De Placido G, Esteves SC, Fischer R, Galliano D, Polyzos NP, Sunkara SK, Ubaldi FM, Humaidan P. A new more detailed stratification of low responders to ovarian stimulation: from a poor ovarian response to a low prognosis concept. Fertil Steril. 2016 Jun;105(6):1452-3. doi: 10.1016/j.fertnstert.2016.02.005. Epub 2016 Feb 26. No abstract available. PMID 26921622
- [Background] Humaidan P, Alviggi C, Fischer R, Esteves SC. The novel POSEIDON stratification of 'Low prognosis patients in Assisted Reproductive Technology' and its proposed marker of successful outcome. F1000Res. 2016 Dec 23;5:2911. doi: 10.12688/f1000research.10382.1. eCollection 2016. PMID 28232864
- [Background] Andersen AN, Devroey P, Arce JC. Clinical outcome following stimulation with highly purified hMG or recombinant FSH in patients undergoing IVF: a randomized assessor-blind controlled trial. Hum Reprod. 2006 Dec;21(12):3217-27. doi: 10.1093/humrep/del284. Epub 2006 Jul 27. PMID 16873892
- [Background] Smitz J, Andersen AN, Devroey P, Arce JC; MERIT Group. Endocrine profile in serum and follicular fluid differs after ovarian stimulation with HP-hMG or recombinant FSH in IVF patients. Hum Reprod. 2007 Mar;22(3):676-87. doi: 10.1093/humrep/del445. Epub 2006 Nov 16. PMID 17110397
- [Background] Vuong TN, Phung HT, Ho MT. Recombinant follicle-stimulating hormone and recombinant luteinizing hormone versus recombinant follicle-stimulating hormone alone during GnRH antagonist ovarian stimulation in patients aged >/=35 years: a randomized controlled trial. Hum Reprod. 2015 May;30(5):1188-95. doi: 10.1093/humrep/dev038. Epub 2015 Mar 3. PMID 25740882
- [Background] Al-Azemi M, Kyrou D, Kolibianakis EM, Humaidan P, Van Vaerenbergh I, Devroey P, Fatemi HM. Elevated progesterone during ovarian stimulation for IVF. Reprod Biomed Online. 2012 Apr;24(4):381-8. doi: 10.1016/j.rbmo.2012.01.010. Epub 2012 Jan 24. PMID 22377153
- [Background] Bungum L, Franssohn F, Bungum M, Humaidan P, Giwercman A. The circadian variation in Anti-Mullerian hormone in patients with polycystic ovary syndrome differs significantly from normally ovulating women. PLoS One. 2013 Sep 4;8(9):e68223. doi: 10.1371/journal.pone.0068223. eCollection 2013. PMID 24023708
- [Background] Gonzalez-Foruria I, Rodriguez I, Martinez F, Rodriguez-Purata J, Montoya P, Rodriguez D, Nicolau J, Coroleu B, Barri PN, Polyzos NP. Clinically significant intra-day variability of serum progesterone levels during the final day of oocyte maturation: a prospective study with repeated measurements. Hum Reprod. 2019 Aug 1;34(8):1551-1558. doi: 10.1093/humrep/dez091. PMID 31334546
- [Background] Griesinger G, Mannaerts B, Andersen CY, Witjes H, Kolibianakis EM, Gordon K. Progesterone elevation does not compromise pregnancy rates in high responders: a pooled analysis of in vitro fertilization patients treated with recombinant follicle-stimulating hormone/gonadotropin-releasing hormone antagonist in six trials. Fertil Steril. 2013 Dec;100(6):1622-8.e1-3. doi: 10.1016/j.fertnstert.2013.08.045. Epub 2013 Sep 29. PMID 24083873
- [Background] Griesinger G, Venetis CA, Tarlatzis B, Kolibianakis EM. To pill or not to pill in GnRH-antagonist cycles: the answer is in the data already! Reprod Biomed Online. 2015 Jul;31(1):6-8. doi: 10.1016/j.rbmo.2015.04.001. Epub 2015 Apr 9. PMID 25985996
- [Background] Golan A, Weissman A. Symposium: Update on prediction and management of OHSS. A modern classification of OHSS. Reprod Biomed Online. 2009 Jul;19(1):28-32. doi: 10.1016/s1472-6483(10)60042-9. PMID 19573287
- [Background] Bosch E, Vidal C, Labarta E, Simon C, Remohi J, Pellicer A. Highly purified hMG versus recombinant FSH in ovarian hyperstimulation with GnRH antagonists--a randomized study. Hum Reprod. 2008 Oct;23(10):2346-51. doi: 10.1093/humrep/den220. Epub 2008 Jun 25. PMID 18583332
- See also: Department of Obstetrics, Gynaecology and Reproduction Hospital Universitari Quirón Dexeus — http://dexeus.com